CLINICAL TRIAL: NCT04574895
Title: Using a Real-Time Risk Prediction Model to Predict Pediatric Venous Thromboembolism Events
Brief Title: Using a Real-Time Risk Prediction Model to Predict Pediatric Venous Thromboembolism (VTE) Events
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Shannon Walker, Clinical Fellow, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 201629
Record Dates: First submitted 2020-09-28; First posted 2020-10-05 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Venous Thromboembolism; Pediatrics; Deep Vein Thrombosis; Pulmonary Embolism
Keywords: Pediatric Hematology; Venous Thromboembolism; Risk Prediction Model; General Pediatrics
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Team biostatistician will remain blinded to the group assignments for performing outcome statistics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VTE risk prediction scores (Other): Patients in the intervention arm will have their VTE risk prediction scores presented to the study team daily on weekdays via an automated report, which will list patients in descending order of risk severity for review by the VTE research team each weekday. Starting with the highest risk patients, the VTE research team will review each patient and clinical situation, and then the VTE research team will directly discuss risks/benefits of prophylactic anticoagulation with the admitting team. Patients with a risk score <2.5% will not be reviewed, and the investigators anticipate most of the intervention arm patients will fall into this category (based on our previous data, the investigators anticipate >90% of all patients will score <2.5%). The VTE risk report will be re-calculated based on updated EHR data every day at midnight.
  Interventions: Other: Hematology Review
- Standard of care (No Intervention): Patients randomized to the control arm will continue to receive current standard of care anticoagulation practice, which is at the discretion of the admitting team. In general, nearly no pediatric patients are offered prophylactic anticoagulation unless a previous VTE has been identified. This currently is at the discretion of the provider and no risk scoring is used. VTE risk prediction scores will be calculated and stored for analysis, these will not be visible to the study team in real time.

INTERVENTIONS:
Other: Hematology Review — VTE study team will review VTE risk percentages provided via automated report daily on weekdays and approach the primary team directly if the patient is appropriate for clinical antithrombotic interventions.
  Arms: VTE risk prediction scores

SUMMARY:
The study will evaluate the effectiveness of a novel, real-time risk prediction model for identifying pediatric patients at risk for developing in-hospital blood clots (or venous thromboembolism [VTE]) based on data easily extracted from the electronic medical record. The study will assess whether using the risk percentages for developing VTE derived from the model increases the number of high-risk patients screened by the pediatric hematology team, which may may lead to an overall reduction in the number of pediatric VTEs seen at Monroe Carell Jr. Children's Hospital at Vanderbilt.

DETAILED DESCRIPTION:
VTE risk factors in adult hospitalized patients are well established and prevention strategies have been implemented for many years. Unfortunately, VTE prevention guidelines are not well established in children, and the pathophysiology of pediatric VTE is sufficiently different from adults that adult studies cannot be extrapolated to pediatrics. There are no randomized trials in pediatrics to determine whether a risk prediction model helps prevent pediatric VTEs.

A risk prediction model was developed that can be applied at admission and updated daily to predict pediatric patients at higher risk for developing a VTE. This model was developed from electronically extracted data from all admissions to the Monroe Carell Jr. Children's Hospital at Vanderbilt from January 1, 2010 to October 31, 2017. Cases were identified based on ICD-9/10 codes. Potential covariates were identified from previous studies and known risk factors for VTE development. The variables with the highest adjusted odds ratio (OR) for developing VTE were history of thrombosis (OR 8.7, 95% confidence interval (CI) 6.6-11.3, p<0.01), presence of a central venous line (OR 4.9, 95%CI 4.0-5.8, p<0.01), and cardiology consultation (OR 4.0, 95%CI 3.3-4.8, p<0.01). Additional significant variables include whether a blood gas was performed, infectious disease consultation, diagnosis of cancer, age, mean corpuscular hemoglobin concentration (MCHC), red cell distribution width (RDW), lactate, and whether surgery was performed.

There have been several smaller pediatric VTE risk prediction models that have been developed and published. However, none of these have been evaluated for efficacy in a prospective trial, and none of these studies have used a randomized trial approach to evaluate benefit in identifying pediatric patients at high risk for developing VTE. Therefore, the investigators are performing a randomized, pragmatic trial to evaluate the pediatric VTE risk prediction model and its efficacy at predicting pediatric patients at higher risk for developing a VTE.

ELIGIBILITY:
Inclusion Criteria:

1. All pediatric patients 0-21 years of age who are admitted to an inpatient unit of Monroe Carell Jr. Children's Hospital at Vanderbilt will be included in the study.

Exclusion Criteria:

1. Receiving prophylactic or therapeutic dosing of anticoagulants, including enoxaparin, warfarin, bivalirudin, apixaban, rivaroxaban, dabigatran, and edoxaban.
2. Patients admitted under "observation status"

Ages: 0 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17427 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Number of VTE Events | 1 year
  Number of VTE events per hospital admission encounter, per study arm. A VTE event will be defined as an acute venous thromboembolic event (e.g. deep vein thrombosis, pulmonary embolism, etc).

SECONDARY OUTCOMES:
Total Number of Patients Started on Anticoagulation | 1 year
  Total number of patients, without contraindications to anticoagulant medications as described by the prescriber information for heparin and enoxaparin determined by the consulting hematologist, who are begun on prophylactic anticoagulation, by study arm
Total Number of High-Risk Patients Started on Anticoagulation | 1 year
  Total number of high-risk patients, without contraindications to anticoagulant medications as described by the prescriber information for heparin and enoxaparin determined by the consulting hematologist, who are begun on prophylactic anticoagulation, by study arm
Total Number of Patients Started On Anticoagulation If It Was Recommended | 1 year
  Total number of patients, without contraindications to anticoagulant medications as described by the prescriber information for heparin and enoxaparin determined by the consulting hematologist, who are begun on anticoagulation medications compared to the total number of patients for which initiation of anticoagulation was recommended by the VTE research team
Total Number of Bleeding Events | 1 year
  Total number of bleeding events per number of patients begun on prophylactic anticoagulation, by study arm, during hospitalization. The bleeding events will be defined and scored using the WHO bleeding scale. Grade 1 (petechial bleeding) and 2 (mild blood loss) will be considered adverse events and grade 3 (bleeding requiring transfusion) and 4 (fatal bleeding) will be considered serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Allison P Wheeler, MD, Study Director — Vanderbilt University Medical Center; Buddy Creech, MD, Study Chair — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Walker SC, Creech CB, Domenico HJ, French B, Byrne DW, Wheeler AP. A Real-time Risk-Prediction Model for Pediatric Venous Thromboembolic Events. Pediatrics. 2021 Jun;147(6):e2020042325. doi: 10.1542/peds.2020-042325. Epub 2021 May 19. PMID 34011634
- [Background] Walker SC, French B, Moore R, Domenico HJ, Wanderer JP, Balla S, Creech CB, Byrne DW, Wheeler AP. Use of a real-time risk-prediction model to identify pediatric patients at risk for thromboembolic events: study protocol for the Children's Likelihood Of Thrombosis (CLOT) trial. Trials. 2022 Oct 22;23(1):901. doi: 10.1186/s13063-022-06823-7. PMID 36273203
- [Result] Walker SC, French B, Moore RP, Domenico HJ, Wanderer JP, Mixon AS, Creech CB, Byrne DW, Wheeler AP. Model-Guided Decision-Making for Thromboprophylaxis and Hospital-Acquired Thromboembolic Events Among Hospitalized Children and Adolescents: The CLOT Randomized Clinical Trial. JAMA Netw Open. 2023 Oct 2;6(10):e2337789. doi: 10.1001/jamanetworkopen.2023.37789. PMID 37831448